CLINICAL TRIAL: NCT00004115
Title: Multicenter Randomized Survival Study of Monoclonal Antibody Radioimmunotherapy: A Multinational Study in Patients With Ovarian Carcinoma Using the HMFG1 Antibody Labeled With 90Yttrium
Brief Title: Monoclonal Antibody Therapy in Treating Patients With Ovarian Cancer or Primary Peritoneal Cancer in Remission Following Surgery and Chemotherapy
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Jonsson Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000067341; UCLA-9712040; ANTISOMA-SMART22; NCI-G99-1604
Record Dates: First submitted 1999-12-10; First posted 2003-01-27 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2003-04

CONDITIONS: Ovarian Cancer; Primary Peritoneal Cavity Cancer
Keywords: stage I ovarian epithelial cancer; stage II ovarian epithelial cancer; stage III ovarian epithelial cancer; stage IV ovarian epithelial cancer; primary peritoneal cavity cancer
MeSH Terms: conditions — Ovarian Neoplasms; Carcinoma, Ovarian Epithelial

INTERVENTIONS:
Radiation: yttrium Y 90 monoclonal antibody HMFG1

SUMMARY:
RATIONALE: Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. It is not yet known whether monoclonal antibody therapy is more effective than observation for ovarian cancer or primary peritoneal cancer that is in remission.

PURPOSE: Randomized phase III trial to compare the effectiveness of monoclonal antibody therapy with that of observation in treating patients who have ovarian cancer or primary peritoneal cancer in remission following surgery and chemotherapy.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the efficacy of yttrium Y 90 monoclonal antibody HMFG1, in terms of survival, in patients with ovarian epithelial carcinoma in remission after debulking surgery and platinum-based chemotherapy.
* Determine the toxicity and tolerability of this treatment regimen in these patients.
* Determine the quality of life of patients treated with this regimen.
* Evaluate this treatment regimen, in terms of the time to relapse, ECOG performance status, frequency of hospitalization, changes in concurrent medication, and incidence and severity of adverse events, in this patient population.

OUTLINE: This is a randomized, parallel, multicenter study. Patients are randomized to one of two treatment arms.

* Arm I: Patients receive standard therapy (observation).
* Arm II: After imaging studies of the peritoneal cavity to verify adequate fluid distribution, patients receive yttrium Y 90 monoclonal antibody HMFG1 intraperitoneally over 1 minute.

Quality of life is assessed in all patients prior to randomization, at weeks 4 and 8, at 3 months, and then every 3 months thereafter.

Patients in arm I are followed at weeks 1, 4, and 8. Patients in arm II are followed weekly for 6 weeks and at weeks 8 and 12. All patients are followed every 3 months for 3 years.

PROJECTED ACCRUAL: A total of 420 patients (210 per treatment arm) will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically proven stage IC, II, III, or IV ovarian epithelial carcinoma or primary peritoneal serous carcinoma
* Prior complete response to 1 platinum-based chemotherapy regimen consisting of at least 5 courses

  * Absence of disease on physical and radiological exam (CT scan/MRI)
  * CA 125 normal
  * No visible evidence of malignant disease on second-look laparoscopy
* No disease relapse even if complete response to a second course of chemotherapy
* Prior bilateral oophorectomy with or without salpingectomy, omentectomy, and total or partial abdominal hysterectomy required
* No known metastases

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 0-2

Life expectancy:

* At least 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Platelet count at least 100,000/mm^3
* Hemoglobin at least 10.0 g/dL

Hepatic:

* SGOT/SGPT no greater than 2 times upper limit of normal

Renal:

* Creatinine no greater than 2.0 mg/dL

Other:

* No other malignancy except basal cell skin cancer
* No serious physical or psychiatric disease that would preclude study entry
* No significant loculation that would preclude good distribution of study medication
* Human antimouse antibody negative

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior murine antibody

Chemotherapy:

* See Disease Characteristics
* No more than 4-8 weeks since prior chemotherapy

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* See Disease Characteristics

Other:

* No concurrent participation in other trials involving adjuvant cancer treatment
* No other concurrent experimental therapies

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-12

CONTACTS AND LOCATIONS:
Overall Officials: Jonathan S. Berek, MD, Study Chair — Jonsson Comprehensive Cancer Center
Locations (1):
- Antisoma, London, England, United Kingdom